CLINICAL TRIAL: NCT00002997
Title: Phase II Trial of Cryoablation for Treatment of Unresectable Colorectal Hepatic Metastases
Brief Title: Cryosurgery in Treating Patients With Unresectable Liver Metastases From Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065545; ECOG-1296
Record Dates: First submitted 1999-11-01; First posted 2004-04-07 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum; liver metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Cryosurgery

INTERVENTIONS:
Procedure: cryosurgery

SUMMARY:
RATIONALE: Cryosurgery for liver metastases may have fewer side effects and improve recovery.

PURPOSE: Phase II trial to study the effectiveness of cryosurgery for patients with unresectable liver metastases from colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the feasibility of conducting a multi-institutional clinical study of cryosurgery for liver metastases. II. Evaluate the morbidity and mortality of cryosurgery for liver metastases when applied in a multi-institutional setting. III. Evaluate the efficacy of cryosurgery for liver metastases as measured by total liver control, local lesion control, and overall survival.

OUTLINE: This is a multi-institutional study. Patients are first confirmed by exploratory laparotomy to have no extrahepatic metastases. They then undergo biopsy of the portal lymph node, after which, full mobilization of liver is recommended. Cholecystectomy is optional but recommended for treatment of tumors adjacent to the gallbladder. After mapping out the location and size of the metastatic tumor by ultrasound, cryoablation of the metastases is carried out. Cryoablation involves the delivery of nitrogen through metallic probes placed surgically into the center of the liver metastases. There are two freeze and thaw cycles for each lesion with synchronous intraoperative ultrasound monitoring of the cryoablation. One centimeter margin of cryoablation is determined by this ultrasound image. Treatment of the liver with regional chemotherapy is not allowed until radiographic and pathologic confirmation of disease progression in the liver. Follow-up is at 3 weeks after surgery and then every 3 months.

PROJECTED ACCRUAL: There will be a maximum of 45 patients accrued in approximately 3 years for this study. This is a two stage accrual design in which 17 patients are first accrued of which 15 should be eligible. If fewer than 11 of the initial 15 eligible patients show no evidence of disease at 3 months, the study stops and treatment is abandoned. If at least 11 patients show no evidence of disease, then 28 additional patients are accrued.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed primary colorectal adenocarcinoma with synchronous and metachronous metastases to liver 1 to 5 liver metastases demonstrated by rapid sequence CT scan or Feridex-enhanced MRI within 2 weeks of registration CT portography not required No single metastasis greater than 6 cm Maximum liver involvement must not be more than 40% by volume No extrahepatic metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Hematopoietic: Platelet count greater than 80,000/mm3 Prothrombin time less than 15.0 seconds Hepatic: Bilirubin less than 2.0 mg/dL Renal: Not specified Other: Must be disease free for at least 5 years except for treated basal cell or squamous cell skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Prior chemotherapy allowed No concurrent regional chemotherapy allowed Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-02-04 (Actual); Primary Completion 2001-01-31 (Actual); Study Completion 2004-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James L. Peacock, MD, Study Chair — James P. Wilmot Cancer Center
Locations (3):
- United States (3):
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of Rochester Cancer Center, Rochester, New York
  - Hahnemann University Hospital, Philadelphia, Pennsylvania